CLINICAL TRIAL: NCT01378130
Title: Central Serous Chorioretinopathy: An Observational Study About Etiology, Course and Prognosis
Brief Title: Central Serous Chorioretinopathy: Etiology, Course and Prognosis
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Sacu, Assoc. Prof. Dr., Medical University of Vienna
Other Study IDs: EK 180/2011
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Central Serous Chorioretinopathy
Keywords: CCS; CSC; Subretinal Fluid; multimodal imaging
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Pathogenesis of central serous chorioretinopathy is not entirely understood yet, therefore further investigations are needed. During this study patients with an acute episode of central serous chorioretinopathy are observed with established ophthalmologic methods (multimodal imagine) every 6 weeks until subretinal fluid is reabsorbed to gain further insides in etiology, course and prognosis of this disease.

DETAILED DESCRIPTION:
Patients with central serous chorioretinopathy are recruited from the Department of Ophthalmology at the Medical University of Vienna. All patients undergo ETDRS visual acuity measurement, Pelli-Robson contrast examination, Amsler-Grid testing, questionnaire testing, ophthalmologic examination, SD-OCT and polarization-sensitive OCT, fundus autofluorescence, fluorescein angiography, indocyanine-green angiography, fundus photo and microperimetry. Patients are re-examined after an interval of 6 weeks until subretinal fluid is entirely reabsorbed to gain further insides in etiology, course and prognosis of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Age over 18 years
* acute episode of Central Serous Chorioretinopathy
* Symptoms for less than two weeks
* no treatment on study eye

Exclusion Criteria:

* bad compliance
* protected patient group (pregnant women)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an acute episode of central serous chorioretinopathy are recruited from the Department of Ophthalmology at the Medical University of Vienna.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Clinical Outcome | 2 years
  OCT, Visus

SECONDARY OUTCOMES:
Subclinical Data | 2 years
  FA findings, retinal sensitivity in Microperimetry, contrast sensitivity, Amsler Grid Test

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Sacu, Ass.Prof.Dr., Principal Investigator — Department of Ophthalmology, Medical University of Vienna, Austria
Locations (1):
- Vienna Gerenal Hospital, Vienna, Austria